CLINICAL TRIAL: NCT01388374
Title: A Study on the (Cost-)Effectiveness of Nurse Practitioners Working at the Primary Out of Hours Emergency Service and the Feasibility of Implementing These Nurses
Brief Title: The (Cost-)Effectiveness of Nurse Practitioners Working at the Primary Out of Hours Emergency Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 80-82800-98-227
Record Dates: First submitted 2011-07-04; First posted 2011-07-06 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Out of Hours Medical Care; Primary Health Care
Keywords: Delivery of Health Care; Nurse Practitioners; Out of Hours Medical Care; Primary Health Care; Emergency Medical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Practitioners Care (No Intervention): Usual medical care provided by a general practitioner at the Primary Out of Hours Emergency Service.
- Nurse Practitioners Care (Experimental): Medical care provided by the Nurse Practitioner at the Primary Out of Hours Emergency Service.
  Interventions: Other: Other, care provided by Nurse Practitioners

INTERVENTIONS:
Other: Other, care provided by Nurse Practitioners — Patients will receive care at the Primary Out of Hours Emergency Service by a Nurse Practitioner instead of a General Practitioner (substitution of care from physicians to nurses).
  Arms: Nurse Practitioners Care

SUMMARY:
The aim of this study is to explore whether the implementation of Nurse Practitioners can lead to a more accessible and efficient patient care at the primary out of hours service.

The primary objectives of the proposed study are:

1. What are the effects of the implementation of NPs on the primary out of hours service in comparison with the current out of hours service? Effects in terms of accessibility, objective and subjective workload of general practitioners, quality of care and patient satisfaction.
2. How efficient is the implementation of NPs in the primary out of hours services?
3. What is the feasibility of the implementation of NPs in the out of hours services? And under which conditions?
4. What are the barriers and facilitating factors considering the implementation of NPs?

DETAILED DESCRIPTION:
The emergency care and primary out of hours care in the Netherlands is under pressure. There is a rising demand from patients for acute care at the primary out of hours service (run by General Practitioners) as well as for the emergency departments (EDs) at the hospitals. The workload for healthcare professionals in these acute care setting is high. Without changes in the organization of primary out of hours care and emergency care, the quality, accessibility and efficiency of the acute care can't be guaranteed in the future.

The substitution of care from General Practitioners (GPs) to Nurse Practitioners (NPs) is seen as one possible solution to decrease the GPs' workload and improve accessibility and efficiency of care without reducing the quality of care.

It turned out that about 80% of the acute complaints is U3 and U4 (low complex and not urgent) and does not necessarily to be seen by a physician.

Based on previous research we expect that the NPs are competent to diagnose and treat almost all low complex and not urgent complaints. During surgery hours (day time) the NPs act in about 90% of the consultations independently.

Hypothetical substitution of care should contribute to enhancing quality, improving accessibility and reducing the workload of doctors. It can also benefit the efficiency of the acute (primary out of hours) care.

However, specific scientific evidence for this is lacking.

In this study we examine whether substitution of care from GPs to NPs in a primary out of hours care setting can contribute to a more accessible and efficient patient care. Also the feasibility of implementing NPs in a primary our of hours setting is examined.

Comparison: Care provided by the Nurse Practitioner will be compared to care provided by a General Practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Patients (with urgency U2, U3, or U4) requesting an appointment at the primary out of hours emergency service during the weekend between 10.00 and 17.00 hours.

Exclusion Criteria (patients seen by a NP):

* Patients under the age of 1 year
* Patients with psychiatric complaints
* Patients with abdominal pain, abdominal infections, chest pain or neck complaints (angina pectoris), headache and dizziness.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12092 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Accessibility of care | 15 months
  Number of patients that have a consult at the Primary Out of Hours Emergency Service; Waiting time; Productivity by NPs in comparison with productivity by GPs.

SECONDARY OUTCOMES:
Quality and safety of care | 15 months
  Quality and safety of care will be measured by video/audio recording. In total, 60 consultations/visits will be recorded. 30 of the General Practitioner and 30 of the Nurse Practitioner. The care between these two disciplines will be compared according to the practice guidelines for General Practitioners (list of indicators).
  Furthermore, we report the amount of adverse events and complications. Also complaints by the patients will be recorded.
Patient satisfaction | 15 months
  Patient satisfaction will be measured by a questionnaire (CQ-index). At baseline and three times during the intervention period questionnaires will be sent to patients who had a consult at the Primary Out of Hours Emergency Service.
Feasibility | 15 months
  Barriers and facilitators will be explored. We collect this information through semi-structured interviews with GPs, practice assistants, NPs and physicians working at the Primary Out of Hours Emergency Service.
Efficiency of care | 15 months
  To measure the efficiency of healthcare, we will measure type of consultation; duration of the consult; type of care provider; number of patients; number of prescriptions; number of test & investigations ordered, referral to other healthcare providers and the emergency department.
  These data will be derived from the electronic medical records and patient questionnaires.
Workload | 15 months
  Objective workload will be measured by the numbers of consults, taking into account the urgency levels of the complaints. This data will be derived from the electronic medical records
  Subjective workload will be measured by a questionnaire. General practitioners as well as the practice assistants at the Primary Out of Hours Emergency Service receive a questionnaire before and after the intervention period to measure satisfaction with care and workload issues
Knowledge/competence of the NPs | 15 months
  After 9 months, we will measure the knowledge of NPs with regard to a number of frequently presented complaints. We will use a 'knowledge test' used to examine the knowledge of GP trainees. Besides NPs also a random selection of GPs (with similar experience of practice) will be invited to fill in the knowledge test.
Cost-analysis | 15 months
  All costs related to care provided by NPs and GPs will be calculated, including number of consultations, resource use, referrals, etc. We will also include the costs for training of GPs and NPs.
  The EQ-D5 will be used as standardized measure for health status of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: M.G.H. Laurant, Dr., Principal Investigator — IQ healthcare, UMC St Radboud
Locations (1):
- Centrale Huisartsen Post (CHP), Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] Bos N et al (2009). Het gebruik van spoedzorg Regio Utrecht 2009. Utrecht: Julius Centrum.
- [Background] Giesen P, et al (2007). Medische zorg buiten kantooruren: de huisartsenpost of de spoedeisende eerste hulp? Huisarts Wet;50(5):202-6.
- [Background] Ministerie van VWS. Beleidsvisie acute zorg. Oktober 2003.
- [Background] VHN (2009). Benchmarkbulletin 2008. Utrecht: VHN.
- [Background] Giesen P, et al (2005). How urgent is the presented morbidity on the GP cooperative? Huisarts Wet; 48: 207-10.
- [Background] De Jongh M & Welling G (2009). Analyse zorgvraag Huisartsenpost Eindhoven. Eindhoven: De Centrale Huisartsenposten Zuidoost Brabant
- [Background] Giesen P, et al (2009). Te snel naar de huisartsenpost. Medisch Cont; 64(6)239-42.
- [Background] IGZ (2004). Spoedeisende hulpverlening; haastige spoed niet overal goed. Den Haag: IGZ
- [Background] Meyboom-de Jong B, van der Kam WJ, Pierik EG, Bosveld HP. [No Friday afternoon peak in the number of patients referred to the emergency room at De Weezenlanden Hospital of Zwolle, May/June 1997]. Ned Tijdschr Geneeskd. 1999 Dec 18;143(51):2562-6. Dutch. PMID 10633796
- [Background] Jaarsma-van Leeuwen I, Hammacher ER, Hirsch R, Janssens M. [Patients without referral treated in the emergency room: patient characteristics and motives]. Ned Tijdschr Geneeskd. 2000 Feb 26;144(9):428-31. Dutch. PMID 10719547
- [Background] van Uden CJ, Winkens RA, Wesseling GJ, Crebolder HF, van Schayck CP. Use of out of hours services: a comparison between two organisations. Emerg Med J. 2003 Mar;20(2):184-7. doi: 10.1136/emj.20.2.184. PMID 12642541
- [Background] van Uden CJ, Crebolder HF. Does setting up out of hours primary care cooperatives outside a hospital reduce demand for emergency care? Emerg Med J. 2004 Nov;21(6):722-3. doi: 10.1136/emj.2004.016071. PMID 15496709
- [Background] RVZ (2003). Acute zorg [Achtergrondstudie].( www.rvz.net )
- [Background] Giesen P, Franssen E, Mokkink H, van den Bosch W, van Vugt A, Grol R. Patients either contacting a general practice cooperative or accident and emergency department out of hours: a comparison. Emerg Med J. 2006 Sep;23(9):731-4. doi: 10.1136/emj.2005.032359. PMID 16921097
- [Background] Jabaaij et al (2006). Diensten de deur uit. Huisartsen verkopen meer ANW-diensten aan een waarnemer. Med Contact; 61 (46): 1840-2.
- [Background] McCarthy ML, Zeger SL, Ding R, Levin SR, Desmond JS, Lee J, Aronsky D. Crowding delays treatment and lengthens emergency department length of stay, even among high-acuity patients. Ann Emerg Med. 2009 Oct;54(4):492-503.e4. doi: 10.1016/j.annemergmed.2009.03.006. Epub 2009 May 6. PMID 19423188
- [Background] Leibowitz R, Day S, Dunt D. A systematic review of the effect of different models of after-hours primary medical care services on clinical outcome, medical workload, and patient and GP satisfaction. Fam Pract. 2003 Jun;20(3):311-7. doi: 10.1093/fampra/cmg313. PMID 12738701
- [Background] Helsloot et al (2006). De eerste schakel. De huisartsgeneeskundige inbreng in de acute zorgketen. Medisch Cont; 61(6): 653-5.
- [Background] Dierick-van Daele AT, Metsemakers JF, Derckx EW, Spreeuwenberg C, Vrijhoef HJ. Nurse practitioners substituting for general practitioners: randomized controlled trial. J Adv Nurs. 2009 Feb;65(2):391-401. doi: 10.1111/j.1365-2648.2008.04888.x. PMID 19191937
- [Background] Dierick-van Daele AT, Steuten LM, Metsemakers JF, Derckx EW, Spreeuwenberg C, Vrijhoef HJ. Economic evaluation of nurse practitioners versus GPs in treating common conditions. Br J Gen Pract. 2010 Jan;60(570):e28-35. doi: 10.3399/bjgp10X482077. PMID 20040165
- [Background] Dierick-van Daele et al (2008). Nurse practitioner in de huisartsenpraktijk: onderzoeksrapport. Maastricht/Eindhoven: UMC Maastricht en Stichting KOH.
- [Background] de Leeuw et al (2009). Taakherschikking in de huisartsenpraktijk: introductie van de Physician Assistant. Utrecht: UMC Utrecht, Julius Centrum voor Gezondheidswetenschappen en Eerstelijns Geneeskunde.
- [Background] Laurant M, Harmsen M, Wollersheim H, Grol R, Faber M, Sibbald B. The impact of nonphysician clinicians: do they improve the quality and cost-effectiveness of health care services? Med Care Res Rev. 2009 Dec;66(6 Suppl):36S-89S. doi: 10.1177/1077558709346277. PMID 19880672
- [Background] Laurant MGH (2007). Changes in skill mix. The impact of adding nurses to the primary care team. [Thesis] Nijmegen: Radboud University Nijmegen.
- [Background] Laurant M, Reeves D, Hermens R, Braspenning J, Grol R, Sibbald B. Substitution of doctors by nurses in primary care. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001271. doi: 10.1002/14651858.CD001271.pub2. PMID 15846614
- [Background] Meulepas MA (2007). Evaluation of a chronic care model for primary care. [Thesis] Nijmegen: Radboud University Nijmegen.
- [Background] Horrocks S, Anderson E, Salisbury C. Systematic review of whether nurse practitioners working in primary care can provide equivalent care to doctors. BMJ. 2002 Apr 6;324(7341):819-23. doi: 10.1136/bmj.324.7341.819. PMID 11934775
- [Background] Hooker (2000). The economic basis of physician assistant practice. Physician Assist; 24: 51-66.
- [Background] Laurant MG, Hermens RP, Braspenning JC, Akkermans RP, Sibbald B, Grol RP. An overview of patients' preference for, and satisfaction with, care provided by general practitioners and nurse practitioners. J Clin Nurs. 2008 Oct;17(20):2690-8. doi: 10.1111/j.1365-2702.2008.02288.x. Epub 2008 Jul 17. PMID 18647199
- [Background] Hollinghurst S, Horrocks S, Anderson E, Salisbury C. Comparing the cost of nurse practitioners and GPs in primary care: modelling economic data from randomised trials. Br J Gen Pract. 2006 Jul;56(528):530-5. PMID 16834880
- [Background] Dierick-van Daele AT, Spreeuwenberg C, Derckx EW, Metsemakers JF, Vrijhoef BJ. Critical appraisal of the literature on economic evaluations of substitution of skills between professionals: a systematic literature review. J Eval Clin Pract. 2008 Aug;14(4):481-92. doi: 10.1111/j.1365-2753.2008.00924.x. Epub 2008 Jul 9. PMID 19126175
- [Background] Vrijhoef B (2002). Effect evaluation of substituting physicians for nurses in the care for chronically ill. Maastricht: University of Maastricht.
- [Background] Miller W, Riehl E, Napier M, Barber K, Dabideen H. Use of physician assistants as surgery/trauma house staff at an American College of Surgeons-verified Level II trauma center. J Trauma. 1998 Feb;44(2):372-6. doi: 10.1097/00005373-199802000-00025. PMID 9498514
- [Background] Schermerhorn et al. (2010). De huisartsenpost te druk? Er gloort licht aan de horizon.... De NP!. Gorinchem: CHP Gorinchem.
- [Background] Burgt R van der, Derckx E, Toemen T (2009). Taakherschikking in de huisartsenzorg: ANW -eindrapport preparatory grant ZonMW-. Eindhoven, Stichting KOH
- [Background] Spenkelink-Schut et al (2009). Training the Physician Assistant in the Netherlands. JEPA; 19 (40): 46-53.
- [Background] Bussemakers et al (2007). De rolverdeling. Taak-herschikking en taakverdeling in de huisartsenpraktijk. Med Contact; 62 (28): 1216-8.
- [Background] Hooker et al (2007). The globalization of the physician assistant profession. Journal of Physician Assistant Education; 18: 76-85.
- [Background] Spenkelink-Schut et al (2006). De Phyisician Assistant. Een niuewe masteropleiding binnen het medisch domein van de gezondheidszorg in Nederland. Vakblad voor opleiding in het gezondheidszorgonderwijs; 5: 18-22.
- [Background] Toemen Th. (2006). Master of ANP-Huisartsenzorg 2004-2006: overzicht inhoud en ICPC-codes modules patiëntenzorg huisarts-geneeskunde. Stichting KOH, Eindhoven.
- [Background] Toemen Th., Ram P. (2006). De NPH-opleiders begeleid -begeleiding van opleiders van nurse practitioners werkzaam in de huisarstenpraktijk. Stichting KOH, Eindhoven.
- [Background] Derckx, EWCC et al (2006). De Nurse Practitioner in de huisartsenpraktijk biedt perspectief! Modern Medicine; 30(3): 103-7.
- [Background] Bruurs et al. Het ijs is gebroken. Eerste ervaringen met physician assistant stemmen hoopvol. Med Contact; 60:443-6.
- [Background] Grol R & Schrijvers AJP (2005). Onderzoeksprogramma Spoedzorg. Nijmegen/Utrecht: Centre for Quality of Care Research/ Julius Centrum
- [Background] Engelen L & Schoonhoven L (2009). Arbeidsmarktproblematiek binnen de spoedzorgketen. Nijmegen: Acute Zorgregio Oost.
- [Background] Derckx & Toemen (2005). Tussen Cure en Care. Nurse Practitioner in de huisartsenpraktijk verdient ichtzelf terug. Med Contact; 60(49):1992-5.
- [Background] Sixma et al (2008). Handboek CQI Ontwikkeling: ricthlijnene en voorschriften voor de ontwikkeling van een CQI meetinstrument (versie 2.0). Utrecht: Centrum Klantervaringen Zorg.
- [Background] Moll van Charante E, Giesen P, Mokkink H, Oort F, Grol R, Klazinga N, Bindels P. Patient satisfaction with large-scale out-of-hours primary health care in The Netherlands: development of a postal questionnaire. Fam Pract. 2006 Aug;23(4):437-43. doi: 10.1093/fampra/cml017. Epub 2006 Apr 26. PMID 16641129
- [Background] Carret ML, Fassa AG, Kawachi I. Demand for emergency health service: factors associated with inappropriate use. BMC Health Serv Res. 2007 Aug 18;7:131. doi: 10.1186/1472-6963-7-131. PMID 17705873
- [Background] Tummers, G. (2002) Workorganisation, work characteristics and their physiological effects on nurses in the Netherlands. International Journal of stressmanagement, 9(3), 183-206.
- [Background] Dale J, Green J, Reid F, Glucksman E. Primary care in the accident and emergency department: I. Prospective identification of patients. BMJ. 1995 Aug 12;311(7002):423-6. doi: 10.1136/bmj.311.7002.423. PMID 7640591
- [Background] Kinnersley P, Anderson E, Parry K, Clement J, Archard L, Turton P, Stainthorpe A, Fraser A, Butler CC, Rogers C. Randomised controlled trial of nurse practitioner versus general practitioner care for patients requesting "same day" consultations in primary care. BMJ. 2000 Apr 15;320(7241):1043-8. doi: 10.1136/bmj.320.7241.1043. PMID 10764366
- [Background] Wensing M, Grol R, Asberg J, van Montfort P, van Weel C, Felling A. Does the health status of chronically ill patients predict their judgements of the quality of general practice care? Qual Life Res. 1997 May;6(4):293-9. doi: 10.1023/a:1018405207552. PMID 9248311
- [Background] Oostenbrink et al (2004). Handleiding voor kostenonderzoek, methoden en richtlijnprijzen voor economische evalauties in de gezondheidszorg. Den Haag
- [Background] Drummond, M. F., O'Brien, B., Stoddart, G. L. & Torrance, G. W. (2003) Methods for the economic evaluation of health care programmes, second edition., Oxford, Oxford University Press.
- [Background] Barber JA, Thompson SG. Analysis and interpretation of cost data in randomised controlled trials: review of published studies. BMJ. 1998 Oct 31;317(7167):1195-200. doi: 10.1136/bmj.317.7167.1195. PMID 9794854
- [Background] Thompson SG, Barber JA. How should cost data in pragmatic randomised trials be analysed? BMJ. 2000 Apr 29;320(7243):1197-200. doi: 10.1136/bmj.320.7243.1197. No abstract available. PMID 10784550
- [Background] Harmsen M, Adang EM, Wolters RJ, van der Wouden JC, Grol RP, Wensing M. Management of childhood urinary tract infections: an economic modeling study. Value Health. 2009 Jun;12(4):466-72. doi: 10.1111/j.1524-4733.2008.00477.x. Epub 2008 Dec 11. PMID 19171007
- [Background] Adang EM, Wensing M. Economic barriers to implementation of innovations in health care: is the long run-short run efficiency discrepancy a paradox? Health Policy. 2008 Dec;88(2-3):236-42. doi: 10.1016/j.healthpol.2008.03.014. Epub 2008 May 8. PMID 18471924
- [Background] Wester F. (1995) Strategieën voor kwalitatief onderzoek. Coutinho 3e druk, Bussum
- [Background] Grol R, Wensing M. (red) Implementatie Effectieve verbetering van de Patiëntenzorg. Maarssen: Elsevier Gezondheidszorg. 3e herziene druk. 2006. ISBN 90 352 2852 9; NUR 882
- [Background] Meulepas M, Laurant M, Derckx E. (2009). Taakherschikking in de huissartsenzorg: POH GGZ als versterking van de eerstelijns GGZ. Modellenwwegwijzer POH GGZ. Eindhoven:Meetpunt Kwaliteit.
- [Background] Derckx, EWCC, vander Burgt M.R, de Bakker D. Vrijhoef HJM (2009): Naar een landelijke implementatie van de NP en de PA in de eerste lijn.Eindhoven: Stichting KOH
- [Derived] Van Der Biezen M, Adang E, Van Der Burgt R, Wensing M, Laurant M. The impact of substituting general practitioners with nurse practitioners on resource use, production and health-care costs during out-of-hours: a quasi-experimental study. BMC Fam Pract. 2016 Sep 13;17(1):132. doi: 10.1186/s12875-016-0528-6. PMID 27619968
- [Derived] Wijers N, Schoonhoven L, Giesen P, Vrijhoef H, van der Burgt R, Mintjes J, Wensing M, Laurant M. The effectiveness of nurse practitioners working at a GP cooperative: a study protocol. BMC Fam Pract. 2012 Aug 7;13:75. doi: 10.1186/1471-2296-13-75. PMID 22870898
- See also: Projectdescription and dutch documentation related to the project — http://www.iqhealthcare.nl/ContentFront/ContentProjects/ProjectsMain.aspx?projectId=411